CLINICAL TRIAL: NCT02955524
Title: Topical Anesthesia to Decrease the Trigeminal-Cardiac Reflex During Intra-arterial Injection of Chemotherapy for Retinoblastoma in Children.
Brief Title: Topical Anesthesia and Intra-arterial Chemotherapy for Retinoblastoma
Acronym: TOPIAC
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: I discontinued this study because I transferred to another institution.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jacqueline L Tutiven, Assistant Professor of Clinical Anesthesiology/Pediatric Anesthesia Dir., University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20161001
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment session 1a (Experimental): Topical ophthalmic anesthesia to participants (#) on each session (letter) of intra-arterial chemotherapy.
  where #1 is the participant identifier and letter-a is the start session with study protocol (most candidates will receive more than 4 sessions in a 6 month period)
  Interventions: Drug: Tetracaine 0.5%; Drug: Lidocaine hydrochloride ophthalmic gel 3.5%

INTERVENTIONS:
Drug: Tetracaine 0.5% — One drop of 0.5% Proparacaine to nasolacrimal Duct to numb the ethmoidal nerve in the nasal passage on the side of the eye to be treated.
Drug: Lidocaine hydrochloride ophthalmic gel 3.5% — 1ml of lidocaine gel is placed over the conjunctivae of the eye to be treated after the patient is under general anesthesia and before the procedure
  Other Names: Akten

SUMMARY:
The objective of this study is to use local topical anesthesia to numb the sensory input, captured by branches of the Trigeminal nerve found on the skin in and around the eye, to decrease a hemodynamic reflex seen during placement of a catheter for intra-arterial chemotherapy (IAC) for eye tumors in children. This Trigeminal-cardiac reflex brings about hemodynamic instability during general anesthesia.

Normally, one could block this sensorial input with ophthalmic peribulbar placement of local anesthetics, but these eyes have malignant growth and invasive procedures may cause more harm. The investigators are aiming to numb the sensory branches of the trigeminal nerve non-invasively and observe for any decrease in these events.

DETAILED DESCRIPTION:
Retinoblastoma is a rare tumor of the eye and accounts for 6% of malignancies in children less than 5 years of age. Pediatric anesthesiologists have observed a series of hemodynamic instability following the insertion of a catheter into the cavernous segment of the internal carotid artery or during manipulation of a micro-catheter into the ophthalmic artery for intra-arterial chemotherapy (IAC) of retinoblastoma cases by neuroradiologists. This reaction has been recently published in case reports and observational studies as the treatment of these tumors have moved into the interventional imaging suites. This reaction closely resembles the "diving reflex" seen when a person is submerged in cold water; known as the trigeminal-cardiac reflex. It manifests as a sudden hemodynamic disturbance in arterial blood pressure, heart rate, arrhythmia and changes in pulmonary compliance.Rescue from a trigeminal-cardiac reflex entails increasing intravascular volume, administrating mild to resuscitative doses of epinephrine and ventilatory support.

Catheter manipulation around the ophthalmic artery can stimulate the afferent pathway of the trigeminal nerve, branches V1 and V2, originating around the eye to be treated.The ethmoidal nerve, from the nasal passage on the same side, is also stimulated. This in turn triggers a response by the vagus nerve with hemodynamic instability.

Method: Participants are placed under general endotracheal anesthesia for this scheduled procedure. One drop of ocular antiseptic (betadine 5%) will be placed in the eye to be treated followed by a drop of topical FDA approved local anesthetic, Tetracaine 0.5%, to the nasolacrimal duct ( inner corner of the eye) on the eye to be treated. This will numb the ethmoidal nerve in the nasal passage. This is followed by 1 ml of 3.5% Lidocaine gel to the surface of the eye. This gel is placed on the surface of the eye and skin around the eye to numb V1 and V2 fibers of the trigeminal nerve. The study will observe if there is any decrease in the intensity of the reflex or incidence of the reflex during placement of the micro-catheter.

ELIGIBILITY:
Inclusion Criteria:

* Children with Retinoblastoma diagnosis scheduled for Intra-arterial chemotherapy under general anesthesia

Exclusion Criteria:

* any candidate with history of allergy to anesthetics or preservatives used in local anesthetics any candidate that has a history of allergic dermatitis any candidate that has an open wound in and around the eye to be treated

Min Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in systolic Blood Pressure | 5 seconds
  Interventionalist will communicate to the investigator of the catheter placement and our outcome measure will be recorded soon after.
Drop in end-tidal C02 | 5 seconds
  Interventionalist will communicate to the investigator of the catheter placement and our outcome measure will be recorded soon after.
Decrease in lung compliance | 5 seconds
  Interventionalist will communicate to the investigator of the catheter placement and our outcome measure will be recorded soon after.
Decrease in oxygen saturation | 5 seconds
  Interventionalist will communicate to the investigator of the catheter placement and our outcome measure will be recorded soon after.
Cardiac arrythmia | 5 seconds
  Interventionalist will communicate to the investigator of the catheter placement and our outcome measure will be recorded soon after.

SECONDARY OUTCOMES:
Recovery from Trigeminal-cardiac event | 2 minutes
  Investigator will communicate when the event is over or rescue drugs given.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Tutiven, MD, Principal Investigator — Director Pediatric Anesthesia Fellowship/Assistant Professor; Norman Halliday, MD, Study Chair — Chief, Pediatric Anesthesiology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scharoun JH, Han JH, Gobin YP. Anesthesia for Ophthalmic Artery Chemosurgery. Anesthesiology. 2017 Jan;126(1):165-172. doi: 10.1097/ALN.0000000000001381. No abstract available. PMID 27748655
- [Result] Jabbour P, Chalouhi N, Tjoumakaris S, Gonzalez LF, Dumont AS, Chitale R, Rosenwasser R, Bianciotto CG, Shields C. Pearls and pitfalls of intraarterial chemotherapy for retinoblastoma. J Neurosurg Pediatr. 2012 Sep;10(3):175-81. doi: 10.3171/2012.5.PEDS1277. Epub 2012 Jul 13. PMID 22793160